CLINICAL TRIAL: NCT00066651
Title: Phase I Study Of SS1(dsFv)-PE38 Anti-Mesothelin Immunotoxin In Advanced Malignancies: I.V. Infusion QOD Dosing
Brief Title: Immunotoxin Therapy in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000316451; NCI-03-C-0243; NCI-6221; NCI-SS1PE-002; NCT00065481 (obsolete NCT alias)
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2006-02

CONDITIONS: Cervical Cancer; Fallopian Tube Cancer; Head and Neck Cancer; Lung Cancer; Malignant Mesothelioma; Ovarian Cancer; Pancreatic Cancer; Primary Peritoneal Cavity Cancer
Keywords: ovarian carcinosarcoma; ovarian clear cell cystadenocarcinoma; ovarian endometrioid adenocarcinoma; ovarian mixed epithelial carcinoma; ovarian serous cystadenocarcinoma; ovarian undifferentiated adenocarcinoma; recurrent ovarian epithelial cancer; Brenner tumor; primary peritoneal cavity cancer; fallopian tube cancer; epithelial mesothelioma; recurrent malignant mesothelioma; recurrent pancreatic cancer; cervical squamous cell carcinoma; recurrent cervical cancer; recurrent non-small cell lung cancer; squamous cell lung cancer; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent metastatic squamous neck cancer with occult primary; recurrent salivary gland cancer; salivary gland squamous cell carcinoma; recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the nasopharynx
MeSH Terms: conditions — Uterine Cervical Neoplasms; Fallopian Tube Neoplasms; Head and Neck Neoplasms; Lung Neoplasms; Mesothelioma, Malignant; Ovarian Neoplasms; Pancreatic Neoplasms; Carcinoma, Ovarian Epithelial; Brenner Tumor; Carcinoma, Non-Small-Cell Lung; Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — SS1(dsFv)PE38

INTERVENTIONS:
Biological: SS1(dsFv)-PE38 immunotoxin

SUMMARY:
RATIONALE: Immunotoxins can locate tumor cells and kill them without harming normal cells. Immunotoxin therapy may be effective in treating advanced solid tumors.

PURPOSE: This phase I trial is studying the side effects and best dose of immunotoxin therapy in treating patients with recurrent unresectable advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of SS1(dsFv)-PE38 immunotoxin in patients with advanced mesothelin-expressing malignancies.

Secondary

* Determine the toxic effects of this drug in these patients.
* Determine the plasma pharmacokinetics of this drug in these patients.
* Determine the response in patients treated with this drug.
* Correlate the induction of antibody against this drug with its pharmacokinetics in these patients.

OUTLINE: This is an open-label, dose-escalation study.

Patients receive a test dose of SS1(dsFv)-PE38 immunotoxin IV over 1-2 minutes on day 1 followed by SS1(dsFv)-PE38 immunotoxin IV over 30 minutes on days 1, 3, and 5. Treatment repeats every 4 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of SS1(dsFv)-PE38 immunotoxin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 3-15 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced malignancy of 1 of the following types:

  * Ovarian cancer

    * All nonmucinous epithelial histologies are eligible
  * Primary peritoneal cavity cancer
  * Fallopian tube cancer
  * Malignant mesothelioma

    * No sarcomatous histology
  * Pancreatic cancer
  * Squamous cell cancer (SCC) of the lung
  * SCC of the cervix
  * SCC of the head and neck
* Recurrent unresectable disease, meeting 1 of the following criteria:

  * Previously treated with definitive standard therapy
  * Patient refused prior standard therapy
* Initial or recurrent tumor positive (at least 30% of tumor cells) for mesothelin by immunohistochemistry* NOTE: *Immunohistochemical evaluation not required for patients with pancreatic cancer
* Measurable or evaluable disease
* No clinically significant pericardial effusion
* No known CNS or spinal cord involvement by tumor

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 75,000/mm^3

Hepatic

* Bilirubin no greater than upper limit of normal (ULN)
* AST and ALT no greater than 2.5 times ULN
* Albumin at least 3.0 g/dL
* Hepatitis B and C negative

  * Seropositive allowed if clinically asymptomatic
* except if clinically asymptomatic and bilirubin and AST and ALT meet the outlined criteria

Renal

* Creatinine no greater than ULN
* Calcium no greater than ULN

Cardiovascular

* No New York Heart Association class II-IV cardiovascular disease

Pulmonary

* Oxygen saturation at least 93% on room air
* DLCO at least 50% of predicted*
* Total lung capacity and vital capacity at least 50% of predicted*
* FEV_1 at least 50% of predicted* NOTE: *For patients with pleural mesothelioma and as clinically indicated

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No infection requiring parenteral antibiotics
* No HIV infection
* Serum neutralizing activity to SS1(dsFv)-PE38 immunotoxin (at 200 ng/mL) no greater than 75%

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* At least 4 weeks since prior therapy and recovered
* No other concurrent antitumor therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-07

CONTACTS AND LOCATIONS:
Overall Officials: Raffit Hassan, MD, Study Chair — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina